CLINICAL TRIAL: NCT06596837
Title: Virtual Reality and Coping with Procedural Pain in Burn Patients
Acronym: VRZPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Zielina (Other)
Collaborators: Vascular surgery, University hospital Královské Vinohrady, Prague (Other); Palacký University, Olomouc (Unknown); VR Space (Unknown)
Responsible Party: Sponsor-Investigator, Martin Zielina, Head of Medical Ethics and Humanities Department, Second Faculty of Medicine, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TL03000090
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Burns; Virtual Reality; Anxiety; Pain
Keywords: Virtual Reality; Pain Reduction; Anxiety; Burn Patients; Presence; Dressing Changes
MeSH Terms: conditions — Burns; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The investigators employed a repeated-measures crossover design. Participants were divided into Experimental: respondents exposed to highly immersive virtual reality (Cold River) or Other: respondents exposed to low-immersive virtual reality (static images) groups based on the sequence of their informed consents: even-numbered participants were assigned to the Other group, and odd-numbered participants to the Experimental group. Each participant attended two consecutive wound care sessions, which consisted of dressing removal, wound cleaning, and the application of new dressings. The investigators incorporated virtual reality (VR) into one segment of each session: either during the initial phase (dressing removal) or the concluding phase (wound cleaning and new dressing application). In their subsequent sessions, participants experienced VR during the segment opposite to their initial session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- respondents exposed to highly immersive virtual reality (Cold River) (Experimental): The experimental group will have a virtual reality (VR) application Cold River in the VR headset that will significantly enhance the sense of immersion (e.g., realistic environment, interactive capabilities) during one part of the dressing change.
  Interventions: Device: virtual reality
- respondents exposed to low-immersive virtual reality (static images) (Other): The control group will have only static images of a snowy landscape in the virtual reality headset during one part of the dressing change.
  Interventions: Device: virtual reality
- Changing dressings without the use of virtual reality (No Intervention): In the study, each dressing change, whether in the experimental or control group, will include a part where the participant will not wear a virtual reality (VR) headset. Each participant will have two different sessions, and the part of the dressing change without the VR headset will occur at a different stage of the change in each session.

INTERVENTIONS:
Device: virtual reality — The investigators manipulated the following two variables within the experimental design:
  Immersion in the virtual environment. This was a nominal variable with two levels: a low-immersive environment (Other group) and a highly immersive environment (Experimental group) using the Cold River application.
  Order of virtual reality (VR) deployment during the first session. This was also a nominal variable with two levels: VR during the first part of the dressing change (removing the dressing) and VR during the second part of the dressing change (cleaning the wound and applying a new dressing). In each subsequent session, the order of VR deployment was swapped for each participant.
  The values of both variables were assigned to participants according to their numbers (e.g., 1. highly immersive, VR first; 2. low immersive, VR first; 3. highly immersive, VR last; 4. low immersive, VR last, etc.).
  Arms: respondents exposed to highly immersive virtual reality (Cold River); respondents exposed to low-immersive virtual reality (static images)

SUMMARY:
The main aim of the project is to reduce the feeling of procedural pain (when changing bandages) in burn patients through a developed and pilot-verified application for virtual reality (hereinafter VR). The first study on this topic was conducted in the US on two pediatric patients. In addition to pharmacological pain therapy, there are a number of non-pharmacological options (eg, relaxation techniques) that are based on distracting attention from the feeling of pain. VR appears to be the most promising of these options and, in addition to distraction, it also reduces anxiety and depressive symptoms and enhances patient cooperation. The studies also agree on the beneficial role of immersivity; a sense of immersion in VR.

DETAILED DESCRIPTION:
The project was preceded by a pilot verification to select an appropriate approach for implementing the research design, including the development of a new VR application that took into account current technological advancements in this field. As part of the pilot verification, a custom application was created based on experiences with existing VR applications designed for therapeutic purposes for burn trauma patients in collaboration with Space s.r.o. Patients meeting the selection criteria (e.g., extent of burns, consent to participate in the study, and other relevant factors) were included in the study after the second dressing change in the dressing room. It was during these dressing changes that procedural pain occurred, first during the removal of old dressings and then during the removal of necrotic tissue and the application of new dressings. Each of these painful procedures was divided into two parts: 1) removal of old dressings; 2) removal of necrotic tissue and application of new dressings. In the study, pain sensation was repeatedly measured using the NPRS (Numeric Pain Rating Scale) and BSPAS (Burns Specific Pain Anxiety Scale) for both parts in at least 30 patients. Before each dressing change, it was randomly determined whether the VR would be used during the first part (removal of old dressings) or only during the second part (removal of necrotic tissue and application of new dressings). Additionally, the part involving VR was further assessed using a short immersion inventory, the Igroup Presence Questionnaire (IPQ). In the end, it was possible to evaluate the effect of VR on pain management during dressing changes in patients with burn trauma. The investigators will continue to measure several variables. The feeling of nausea will be assessed in a virtual environment on an ordinal scale from 0, indicating no nausea, to 10, indicating the worst imaginable nausea. Age will be recorded and categorized into six ordinal groups ranging from 18 to 70 years and older. The type of medications participants are currently taking will be recorded, categorized into six levels, including options ranging from none to five types of medications, such as strong opioids and analgesics. The total body surface area (TBSA) burned will be measured, with categories ranging from 0.4% to 45% or more. Additionally, the investigators will assess how the burn was caused, with categories including electro trauma, scalding, chemical trauma, frostbite, and flame burns. They will also evaluate participants' gaming and VR experience, determining whether participants consider themselves gamers, play games regularly, or have personal experience with virtual reality. These measurements aim to provide a detailed understanding of the participants´ conditions and their responses during the study.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a thermal injury covering a total body surface area of 0.4% or more
* Actively receiving therapy for the injury
* Proficient in the Czech language

Exclusion Criteria:

* Presence of facial burns
* Acute psychotic illness
* Neurodegenerative diseases
* Other neurological conditions associated with potential cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Pain Change During Dressing Changes - VR vs. Non-VR Phases | From the first dressing change in the study to the second change within one week.
  NPRS (Numeric Pain Rating Scale) We measured the intensity of the pain. The eleven levels of this ordinal variable: are from 0 (not at all) to 10 (the worst I can imagine).
Anxiety Change During Dressing Changes - VR vs. Non-VR Phases | From the first dressing change in the study to the second change within one week.
  BSPAS (Burn Specific Pain Anxiety Scale) We measured pain-related and anticipatory anxiety. The eleven levels of this ordinal variable have nine items: from 0 (not at all) to 10 (the worst I can imagine), ranging from 0 to 90. The higher, the worse.
Presence Change During Dressing Changes - VR vs. Non-VR Phases | From the first dressing change in the study to the second change within one week.
  IPQ (Igroup Presence Questionnaire) We measured the sense of presence experienced in a virtual environment. The seven levels of this ordinal variable have fourteen items. The IPQ measures overall presence (General Presence), ranging from 0 to 7, and three distinct components: Spatial Presence (ranging from 0 to 35), Involvement (ranging from 0 to 28), and Realism (ranging from 0 to 28). Each scale ranges from 0 to 7.
Nausea Change During Dressing Changes - VR vs. Non-VR Phases | From the first dressing change in the study to the second change within one week.
  Nausea We measured nausea in a virtual environment. The eleven levels of this ordinal variable are: from 0 (not at all) to 10 (the worst I can imagine).

SECONDARY OUTCOMES:
Participant demographics (SEX) | From the first dressing change in the study to the second change within one week.
  SEX We measured sex of participants. This nominal, binary variable has two levels: 0 (woman) and 1 (man).
Participant demographics (AGE) | From the first dressing change in the study to the second change within one week.
  AGE We measured the age of participants. This ordinal variable has six levels: 18 to 28, 29 to 39, 40 to 48, 49 to 59, 60 to 69, 70 and over.
Participant demographics (EDUCATION) | From the first dressing change in the study to the second change within one week.
  EDUCATION We measured highest level of education of participants. This nominal variable has three levels: primary school, secondary school, higher education.
Burn characteristics (HOW THE BURN WAS CAUSED) | From the first dressing change in the study to the second change within one week.
  HOW THE BURN WAS CAUSED We measured how the burn was caused. This nominal variable has six levels : Electro trauma, scalding, chemical trauma, frostbite, flame burns and others.
Burn characteristics (TBSA) | From the first dressing change in the study to the second change within one week.
  TBSA We measured the Total Body Surface Area (TBSA) burned. This categorical variable is divided into ten levels: 0.4% to 4.99%, 5% to 9.99%, 10% to 14.99%, 15% to 19.99%, 20% to 24.99%, 25% to 29.99%, 30% to 34.99%, 35% to 39.99%, 40% to 44.99%, and 45% or more.
Burn characteristics (LOCATION OF THE BURN) | From the first dressing change in the study to the second change within one week.
  We measured location of the burn. The levels of this nominal variable correspond to any part of the body, based on the Lund and Browder (LB) chart.

OTHER OUTCOMES:
CURRENT MEDICATION | From the first dressing change in the study to the second change within one week.
  We measured what medications participants were currently taking. This nominal variable has six levels: none to five types of medication (strong opioids, analgesics, anticonvulsants, antidepressants, and benzodiazepines).
GAME PLAYING EXPERIENCE | From the first dressing change in the study to the second change within one week.
  We measured gamer playing experience. This nominal, binary variable has three items: yes and no (Do you consider yourself a computer gamer?, Do you play computer games regularly?, Have you played computer games regularly in the last 6 months?).
VR EXPERIENCE | From the first dressing change in the study to the second change within one week.
  We measured VR experience. This nominal, binary variable has two items: yes and no (Do you have personal experience with virtual reality?, Do you regularly use virtual reality for gaming or work?).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zielina, Dr., Principal Investigator — Charles University, Czech Republic
Locations (1):
- Prague Burn Center, University Hospital Královské Vinohrady, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: start date: September 30, 2024 end date: September 30, 2029
Access Criteria: The anonymized dataset is accessible on the Open Science Framework (OSF) at https://osf.io/embrj/?view_only=5a74f28a0bee4c388d415596bf159bad and can also be requested via martin.zielina@lfmotol.cuni.cz.
URL: https://osf.io/embrj/?view_only=5a74f28a0bee4c388d415596bf159bad

REFERENCES:
- See also: OSF pre-registration — https://osf.io/gmv79